CLINICAL TRIAL: NCT06401408
Title: Effect of Virtual Reality Headsets on Pain, Anxiety, Fear and Physiological Parameters in Children Who Had Skin Prick Test Applied
Brief Title: Effect of Virtual Reality Headsets on Fear Anxiety and Physiological Parameter in Skin Prick Test
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kazım Bagci, Clinical nurse specialist, TC Erciyes University
Other Study IDs: ERU-NF-KB-01
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Allergy
Keywords: allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: Before starting the skin prick test, the child and his/her family who meet the inclusion criteria of the study will be informed about the use of virtual reality headsets(VRH) and volunteer consent forms will be obtained. Before starting the test, the Introductory Characteristics Form for Children and Their Families and scales will be applied to the children and the child's physiological parameters will be taken. Then, the children will be fitted with an VRH and watched an animated film determined in line with the child's age group, developmental characteristics and expert opinions.After the child starts watching the video, skin prick test procedures will be initiated and the child will be allowed to watch the video until the test ends. After the test is completed, physiological parameters will be taken again and scales will be applied.
- control group: No intervention/application will be performed on the children who will be included in the control group. The Introductory Characteristics of Children and Their Families Form and scales will be administered to the children in the control group simultaneously with the experimental group (in the form of pretest-posttest). Additionally, physiological parameters will be taken simultaneously with the experimental group.

SUMMARY:
The goal of this clinical trial is determine the effect of virtual reality headsets on pain, anxiety, fear and physiological parameters in children aged 4-7 years who undergoing skin prick test. The main questions it amis to answer are:

Virtual reality headsets effect on the pain that during the procedure

Virtual reality headsets effect on the anxiety that occurs during the procedure

Virtual reality headsets effect on the fear that occurs during the procedure

Virtual reality headsets effect on physiological parameters (heart rate, blood pressure, respiratory rate) during the procedure

DETAILED DESCRIPTION:
Before starting the skin prick test, the child and his/her family who meet the inclusion criteria of the study will be informed about the use of virtual reality headsets(VRH) and volunteer consent forms will be obtained. Before starting the test (5 minutes before), the Introductory Characteristics Form for Children and Their Families and scales (so that the pain, fear and anxiety scores predicted by the children before the procedure will be measured) will be applied to the children and the child's physiological parameters (heart rate, blood pressure, respiratory rate, oxygen saturation value) will be taken. Then, the children will be fitted with an VRH and watched an animated film (approximately 15 minutes long) determined in line with the child's age group, developmental characteristics and expert opinions.After the child starts watching the video, skin prick test procedures will be initiated and the child will be allowed to watch the video until the test ends. After the test is completed (5 minutes later), physiological parameters will be taken again and scales (thus measuring the pain, fear and anxiety scores felt by the children during the procedure) will be applied.

Control group application phase:

No intervention/application will be performed on the children who will be included in the control group. The Introductory Characteristics of Children and Their Families Form and scales will be administered to the children in the control group simultaneously with the experimental group (in the form of pretest-posttest). Additionally, physiological parameters will be taken simultaneously with the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 4-7,
2. Does not have a chronic or genetic disease,
3. No mental, visual or hearing impairment,
4. No analgesics or sedatives were administered at least one hour before the test procedure,
5. Both he and his parents are open to communication and cooperation,
6. Children who both themselves and their parents volunteer to participate in the research and give verbal and written consent will be included.

Exclusion Criteria:

1. Those who are outside the 4-7 age range,
2. Having a chronic or genetic disease,
3. Mentally, visually or hearing impaired,
4. Applying analgesics and sedatives at least one hour before the test procedure,
5. The child who cannot adapt to virtual reality glasses,
6. Both he and his parents do not cooperate,
7. Children who neither they nor their parents volunteer to participate in the research and who do not give verbal or written consent will not be included in the research.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population of the study will consist of children aged 4-7 years who underwent skin prick test between September 01, 2023 and March 01, 2024 in the Pediatric Allergy Outpatient Clinic of Erciyes University Health Application and Research Center Fevzi Mercan-Mustafa Eraslan Children's Hospital. In the power analysis (effect size= 1.32 α= 0.05, β= 0.95) performed in GPower 3.1 with the findings of the study by Stassart and Giebels (2022), the sample size was determined as experimental (SGG) group=16 and control group=16. At the end of the study, power analysis will be calculated using pain scores and it will be decided whether the sample size is sufficient or not.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Children's Fear Scale (CFS) | 4 weeks
  To conduct an initial investigation of the psychometric properties of the Children's Fear Scale (CFS; based on the adult Faces Anxiety Scale) with young school-age children.The Child Fear Scale (CFS) developed by McMurtry et al. is used to assess the fear levels of children aged 4-10 years. In the scale, 5 cartoon face pictures are used. Anxiety level is evaluated with numbers between "0" and "4". A score of "0" indicates "no anxiety" and a score of "4" indicates "severe anxiety". The validity and reliability of the scale was conducted by Ozalp-Gerceker et al. in 2018. The content validity index is 0.89.Support was found for interrater reliability and test retest reliability of the CFS for measuring children's fear during venipuncture.

SECONDARY OUTCOMES:
Children's Anxiety Meter-State (CAM-S) | 4 weeks
  The CAM scale is drawn to resemble a thermometer with a bulb at the bottom and horizontal lines at intervals going up to the top. Children are instructed to "Pretend that all of your worried or nervous feelings are in the bulb or bottom part of the thermometer. If you are a little bit worried or nervous, the feelings might come up in the thermometer just a little bit.Put a line on the thermometer showing how much worry or nervousness you feel."When children did not understand this analogy, we used an alternate script that did not explicitly describe a thermometer. Children were asked to "Pretend that all of your worried or nervous feelings are in the very bottom down here. If you are a little bit worried or nervous, the feelings might come up just a little bit. If you are very, very worried or nervous, the feelings might go all the way to the top. Put a line showing how much worry or nervousness you feel."

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Tahan, Prof. Dr., Study Chair — responsible for medical procedures
Locations (1):
- Erciyes University Health Application and Research Center Fevzi Mercan-Mustafa Eraslan Children's Hospital, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Result] Ersig AL, Kleiber C, McCarthy AM, Hanrahan K. Validation of a clinically useful measure of children's state anxiety before medical procedures. J Spec Pediatr Nurs. 2013 Oct;18(4):311-9. doi: 10.1111/jspn.12042. Epub 2013 Jun 25. PMID 24094126
- [Result] Addab S, Hamdy R, Thorstad K, Le May S, Tsimicalis A. Use of virtual reality in managing paediatric procedural pain and anxiety: An integrative literature review. J Clin Nurs. 2022 Nov;31(21-22):3032-3059. doi: 10.1111/jocn.16217. Epub 2022 Jan 23. PMID 35068011
- [Result] Antunes J, Borrego L, Romeira A, Pinto P. Skin prick tests and allergy diagnosis. Allergol Immunopathol (Madr). 2009 May-Jun;37(3):155-64. doi: 10.1016/S0301-0546(09)71728-8. Epub 2009 Jul 23. PMID 19769849
- [Result] Barni S, Liccioli G, Sarti L, Giovannini M, Novembre E, Mori F. Immunoglobulin E (IgE)-Mediated Food Allergy in Children: Epidemiology, Pathogenesis, Diagnosis, Prevention, and Management. Medicina (Kaunas). 2020 Mar 4;56(3):111. doi: 10.3390/medicina56030111. PMID 32143431
- [Result] Backer V, Nolte H, Pedersen L, Dam N, Harving H. Unawareness and undertreatment of asthma: follow-up in a different geographic area in Denmark. Allergy. 2009 Aug;64(8):1179-84. doi: 10.1111/j.1398-9995.2009.01994.x. Epub 2009 Feb 20. PMID 19243364
- [Result] Bodtger U, Jacobsen CR, Poulsen LK, Malling HJ. Long-term repeatability of the skin prick test is high when supported by history or allergen-sensitivity tests: a prospective clinical study. Allergy. 2003 Nov;58(11):1180-6. doi: 10.1046/j.1398-9995.2003.00323.x. PMID 14616131
- [Result] Chan E, Foster S, Sambell R, Leong P. Clinical efficacy of virtual reality for acute procedural pain management: A systematic review and meta-analysis. PLoS One. 2018 Jul 27;13(7):e0200987. doi: 10.1371/journal.pone.0200987. eCollection 2018. PMID 30052655
- [Result] Cheng Z, Yu S, Zhang W, Liu X, Shen Y, Weng H. Virtual reality for pain and anxiety of pediatric oncology patients: A systematic review and meta-analysis. Asia Pac J Oncol Nurs. 2022 Sep 28;9(12):100152. doi: 10.1016/j.apjon.2022.100152. eCollection 2022 Dec. PMID 36389624